CLINICAL TRIAL: NCT04112446
Title: A Phase I, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Saroglitazar Following a Single Oral Dose of [14C]-Saroglitazar Magnesium in Healthy Male Subjects
Brief Title: Study to Evaluate Absorption, Metabolism and Excretion of Single-dose [14C]-Saroglitazar in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SARO.19.002
Record Dates: First submitted 2019-09-11; First posted 2019-10-02 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — saroglitazar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): 4 mg [14C]-saroglitazar magnesium (approximately 100 μCi) oral suspension
  Interventions: Drug: Saroglitazar magnesium

INTERVENTIONS:
Drug: Saroglitazar magnesium — On Day 1, subjects will receive a single oral dose of [14C]-saroglitazar magnesium
  Other Names: not any

SUMMARY:
This will be a Phase I, open-label, nonrandomized, single-dose study in healthy male subjects.

DETAILED DESCRIPTION:
Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the dose administration. Subjects will be admitted into the Clinical Research Unit (CRU) on Day -1 and be confined to the CRU until at least Day 8. On Day 1, subjects will receive a single oral dose of [14C]-saroglitazar magnesium. Subjects will be discharged if the following discharge criteria are met: plasma radioactivity levels below the limit of quantitation for 2 consecutive collections and ≥ 90% mass balance recovery, or ≤ 1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 3 consecutive 24-hour periods in which both are collected. If discharge criteria are not met by Day 8, subjects will remain in the CRU up to Day 12.

ELIGIBILITY:
Inclusion Criteria:

1. Males, of any race, between 18 and 55 years of age, inclusive.
2. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and/or Check-in as assessed by the Investigator (or designee).
4. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
5. History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. Known hypersensitivity to either saroglitazar magnesium or other PPAR agonists, and/or the excipients in the saroglitazar magnesium formulation.
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). History of cholecystectomy will not be allowed.
5. Subjects with congenital nonhemolytic hyperbilirubinemia (eg, suspicion of Gilbert's syndrome based on total and direct bilirubin).
6. History of alcoholism or drug/chemical abuse within 1 year prior to Check-in.
7. Alcohol consumption of > 14 units per week. One unit of alcohol equals 12 oz (360 mL) of beer, 1½ oz (45 mL) of liquor, or 5 oz (150 mL) of wine.
8. Positive urine drug screen at Screening or positive alcohol breath test result or positive urine drug screen at Check-in.
9. Positive hepatitis panel and/or positive human immunodeficiency virus test ( Appendix 2).
10. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing or 5 times the t1/2 (whichever is longer).
11. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
12. Use or intend to use any prescription medications/products within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
13. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
14. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
15. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in, or positive cotinine at Screening or Check-in.
16. Receipt of blood products within 2 months prior to Check-in.
17. Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
18. Poor peripheral venous access.
19. Have previously completed or withdrawn from this study or any other study investigating saroglitazar magnesium, and have previously received the investigational product.
20. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.
21. Subjects who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 4 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study. The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the Code of Federal Regulations (CFR) recommended levels considered safe, per United States (US) Title 21 CFR 361.1: less than 5,000 mrem whole-body annual exposure with consideration given to the half-lives of the previous radiolabeled study drugs received.
22. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
AUC from time zero to infinity (AUC0-∞) | At predose to maximum up to Day 12
  Area under the time curve from time zero to infinity will be calculated for saroglitazar and saroglitazar sulfoxide in plasma, and total radioactivity in whole blood and plasma
AUC from time zero to the last quantifiable concentration (AUC0-t) administration of [14C]-saroglitazar magnesium | At predose to maximum up to Day 12
  Area under the time curve from time zero to the last quantifiable concentration will be calculated for saroglitazar and saroglitazar sulfoxide in plasma, and total radioactivity in whole blood and plasma
Cmax | At predose to maximum up to Day 12
  Maximum observed concentration will be calculated for saroglitazar and saroglitazar sulfoxide in plasma, and total radioactivity in whole blood and plasma
Tmax | At predose to maximum up to Day 12
  Time to reach maximum observed concentration will be calculated for saroglitazar and saroglitazar sulfoxide in plasma, and total radioactivity in whole blood and plasma
t1/2 | At predose to maximum up to Day 12
  Apparent terminal elimination half-life will be calculated for saroglitazar and saroglitazar sulfoxide in plasma, and total radioactivity in whole blood and plasma
Apparent total clearance (CL/F) | At predose to maximum up to Day 12
  The apparent total clearance (CL/F) will be determined for saroglitazar
Apparent volume of distribution (Vz/F) during the terminal elimination phase | At predose to maximum up to Day 12
  The Apparent volume of distribution (Vz/F) during the terminal elimination phase will be determined for saroglitazar
AUC0-∞ of plasma saroglitazar relative to AUC0-∞ of plasma total radioactivity (AUC0-∞ Plasma saroglitazar/Total Radioactivity Ratio) | At predose to maximum up to Day 12
  AUC0-∞ of plasma saroglitazar relative to AUC0-∞ of plasma total radioactivity (AUC0-∞ Plasma saroglitazar/Total Radioactivity Ratio) will be calculated
AUC0-∞ of whole blood total radioactivity to AUC0-∞ of plasma total radioactivity (AUC0 ∞ Blood/Plasma Ratio) | At predose to maximum up to Day 12
  AUC0-∞ of whole blood total radioactivity to AUC0-∞ of plasma total radioactivity (AUC0 ∞ Blood/Plasma Ratio) will be calculated
Mean residence time | At predose to maximum up to Day 12
  Mean residence time for saroglitazar and saroglitazar sulfoxide will be calculated
Total radioactivity amount excreted in urine and feces | At predose to maximum up to Day 12
  Amount of radioactivity excreted in urine and Feces will be calculated.
Percentage radioactivity excreted in urine and feces | At predose to maximum up to Day 12
  Percentage radioactivity excreted in urine and Feces will be calculated.
Renal clearance (CLR) | At predose to maximum up to Day 12
  Renal clearance for saroglitazar and saroglitazar sulfoxide will be determined

SECONDARY OUTCOMES:
Metabolic profile/ identifications of metabolites and probable structure elucidation for saroglitazar in plasma, urine, and feces | Maximum up to Day 12
  Metabolic profile/ identifications of metabolites and probable structure elucidation for saroglitazar in different matrices like plasma, urine, and feces will be performed and reported
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Maximum up to Day 12
  Incidence and severity of AEs as a measure of safety and tolerability will be measured and reported

OTHER OUTCOMES:
Amount of Saroglitazar excreted in feces | At predose to maximum up to Day 12
  Amount of Saroglitazar in Fecal samples will be calculated.
Percentage of Saroglitazar excreted in feces | At predose to maximum up to Day 12
  Percentage of Saroglitazar excreted in Fecal samples will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: John E. Blanchard, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States